CLINICAL TRIAL: NCT00754403
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Effects on Glycemic Control With Concomitantly Administered Pioglitazone HCl and Metformin HCl Extended Release (Fortamet®) in Subjects With Type 2 Diabetes
Brief Title: Efficacy of Pioglitazone and Fortamet Combination Therapy in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-OPIXT-010; U1111-1114-2423 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 30 mg QD + Metformin 1000 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and metformin
- Metformin 1000 mg QD (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone and metformin — Pioglitazone 30 mg, tablets, orally, once daily and metformin 1000 mg, tablets, orally once daily for up to 16 weeks.
  Other Names: Actos; AD-4833XT; Fortamet
  Arms: Pioglitazone 30 mg QD + Metformin 1000 mg QD
Drug: Metformin — Pioglitazone placebo-matching tablets, orally, once daily and metformin 1000 mg, tablets, orally once daily for up to 16 weeks.
  Other Names: Fortamet
  Arms: Metformin 1000 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy of pioglitazone and metformin combination therapy, once daily (QD), on glycosylated hemoglobin in adults with type 2 diabetes.

DETAILED DESCRIPTION:
Pioglitazone (ACTOS®) is a member of a class of oral antidiabetic agents known as thiazolidinediones. The insulin-sensitizing actions of thiazolidinediones are at least partially mediated through the peroxisome proliferator-activated receptor gamma. These receptors are found primarily in adipocytes, vascular endothelial cells, monocytes, hepatocytes, and to a lesser extent myocytes.

Metformin was developed as an extended-release formulation of metformin hydrochloride and designed for once-a-day oral administration. Metformin is an antihyperglycemic agent, which improves glucose tolerance in patients with, type 2 diabetes, lowering both basal and postprandial plasma glucose.

On 15 July 1999, the FDA approved pioglitazone for use as an adjunct to diet and exercise to improve glycemic control in patients with type 2 diabetes. Pioglitazone is indicated for monotherapy and for use in combination with sulfonylureas, metformin, or insulin when diet and exercise plus the single agent do not result in adequate glycemic control. On 26 November 2003, the FDA approved the combined use of pioglitazone with metformin.

This study is designed to evaluate the effect on glycemic control when pioglitazone and metformin are taken together. Individuals participating in this study will provide written informed consent and will be required to commit to a screening visit and approximately 5 additional visits at the study center. Study participation is anticipated to be about 31 weeks (or approximately 8 months). Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study
* Diagnosed with type 2 diabetes and must have received appropriate counseling on lifestyle modification for type 2 diabetes including diet and exercise.
* If taking metformin monotherapy or metformin and sulfonylurea combination therapy, has a glycosylated hemoglobin greater than or equal to 7.5% and less than or equal to 9.0% at screening and randomization.
* If naïve or taking sulfonylurea monotherapy has an glycosylated hemoglobin greater than or equal to 8.5% and less than or equal to 10.0% at screening and greater than or equal to 7.5% and less than or equal to 9.0% at randomization.

Exclusion Criteria

* Has type 1 diabetes mellitus
* Currently taking any thiazolidinedione or have taken any thiazolidinedione within 12 weeks prior to screening
* Has congestive heart failure; has a triglyceride level greater than 500 mg per dL
* Diastolic blood pressure greater than 100 mmHg or a systolic pressure greater than 160 mmHg
* Body mass index greater than or equal to 42 kg/m2 (weight /height2)
* Alanine transaminase level greater than or equal to 2.5 times the upper limit of normal, active liver disease, or jaundice.
* Male subjects who have a serum creatinine level greater than or equal to 1.5 mg per dL; female subjects who have a serum creatinine level greater than or equal to 1.4 mg per dL at the screening visit and at randomization.
* Currently using insulin or has used insulin 3 months prior to Screening
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Chronically used oral or parenteral glucocorticoids (eg, prednisone, cortisone, hydrocortisone, dexamethasone)
  * Niacin greater than 200 mg per day, including niacin-containing products such as Advicor - 3 months prior to screening and during the study
  * Chronically used steroid-joint injections - 3 months prior to screening and during the study
  * Thiazolidinediones - 3 months prior to screening and during the study
  * Insulin - 3 months prior to screening
  * Other oral antidiabetic medications (eg, nateglinide [Starlix], acarbose [Precose]) with the exception of sulfonylurea - 3 months prior to screening and during the study
  * Metformin - Fortamet Stabilization and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from randomization in Glycosylated Hemoglobin | Final Visit

SECONDARY OUTCOMES:
Change from randomization in Fasting Plasma Glucose | Final Visit
Change from randomization in Insulin | Final Visit
Change from randomization in Pro-Insulin | Final Visit
Change from randomization in Homeostasis Model Assessment | Final Visit
Change from randomization in Triglycerides | Final Visit
Change from randomization in Total Cholesterol | Final Visit
Change from randomization in Low-Density Lipoprotein Cholesterol | Final Visit
Change from randomization in high-density Lipoprotein Cholesterol | Final Visit
Change from randomization in Lipid Fractionation | Final Visit
Change from randomization in High Sensitivity C-Reactive Protein | Final Visit
Change from randomization in Creatine Phosphokinase | Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI